CLINICAL TRIAL: NCT02848911
Title: A Phase I Dose-escalation Study to Assess the Safety of AFM11 (CD19 x CD3 TandAb®) in Patients With Relapsed or Refractory Adult B-precursor Acute Lymphoblastic Leukemia
Brief Title: Safety Study to Assess AFM11 in Patients With Relapsed or Refractory Adult B-precursor ALL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision was made to terminate the AFM11 development
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFM11-102
Record Dates: First submitted 2016-07-18; First posted 2016-07-29 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Leukemia, B-Cell
Keywords: acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFM11 (Experimental): IV (intravenous) infusion, dose escalation
  Interventions: Drug: AFM11

INTERVENTIONS:
Drug: AFM11 — Accelerated-titration dose-escalation with 1 patient per dose-level, followed by standard dose-escalation (3 + 3 design), Treatment duration: 2 weeks

SUMMARY:
The purpose of the study is to determine the maximum tolerated dose (MTD) in patients with acute lymphoblastic leukemia (ALL) and to determine the safety and tolerability of increasing doses and different infusion times of AFM11 infusion in patients with adult B-precursor ALL

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is an aggressive type of leukemia characterized by an overproduction of lymphoblasts or lymphocytes in the bone marrow and the peripheral blood; it is frequently accompanied by suppression of normal hematopoiesis. It can spread to the lymph nodes, spleen, liver, the central nervous system (CNS), and other organs (sanctuary sites). Without treatment, ALL usually progresses quickly.

B- and T-cell lymphoblastic leukemia cells express surface antigens that parallel their respective developmental lineages. Precursor B-cell ALL cells typically express CD10, CD19, and CD34 on their surface, along with nuclear terminal deoxynucleotide transferase. About 20% of adult ALL patients have a cytogenetic abnormality that is indistinguishable from the Philadelphia chromosome (Ph1, t(9;22)), according to the National Cancer Institute (NCI).

The rationale for the use of AFM11 is based on its ability to bind to both malignant cells via its anti-CD19 domain and to T-cells via its anti-CD3 domains. This results in the formation of the "immunological synapse" and the subsequent T-cell activation on leading to killing of malignant cells. AFM11 has 2 binding sites for CD19 and 2 for CD3, its molecular weight is ~ 105kDa compared to diabodies like blinatumomab with one binding site for each target and a much lower molecular weight ~ 55kDa. In addition, preclinical experiments have shown that AFM11 has about a 100 fold higher affinity to CD3 compared to diabodies and is inducing higher cytotoxicity in vitro in the presence of low effector:target cell ratios. These differences might allow for a shortening of the infusion times and potentially higher clinical efficacy compared to blinatumomab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19+ B-precursor Philadelphia-chromosome negative ALL relapsed after at least induction and consolidation or having refractory disease and who are not candidates for bone marrow transplant (including both peripheral blood and hematopoietic stem cell transplant [HSCTs]) with a curative intent at time of screening
2. Patients with CD19+ Philadelphia-chromosome positive ALL who failed or were intolerant to therapy with at least 2 approved tyrosine kinase inhibitors
3. More than 5% blasts in bone marrow
4. In patients with high tumor burden (e.g., more than 50% blasts, or more than 15,000 blasts /µL blood, or elevated lactate dehydrogenase [LDH]) > 2 × upper limit of normal [ULN]), a pre treatment with 10 mg/m2 dexamethasone and 200 mg cyclophosphamide could be administered for up to 5 days.
5. Patients of both genders, age ≥ 18
6. Homogenous CD19 expression on leukemic blasts must be confirmed by either:

   1. Prior results from a CD19+ staining or flow cytometry at the most recent available diagnostic bone marrow biopsy or aspirate, or
   2. Submission of a recent bone marrow biopsy for staining for CD19 positivity. The results of this testing need to be available prior to start of AFM11 treatment.
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. Life expectancy of at least 3 months
9. Ability to understand the patient information and informed consent form
10. Signed and dated written informed consent

Exclusion Criteria:

1. Autologous HSCT within 3 months prior to start of AFM11 treatment
2. Active acute or chronic graft-versus-host disease. All graft-versus-host disease medication should be omitted for at least 4 weeks prior to start of AFM11 treatment.
3. Allogeneic HSCT within 3 months prior to start of AFM11 treatment
4. Prior treatment with blinatumomab or any other CD19 targeting T-cell engager, including CD19 CAR-T cells
5. Treatment with donor-lymphocyte infusions within 4 weeks of start of AFM11 treatment or existing Graft versus Host Disease (GvHD)
6. Known or suspected central nervous system (CNS) involvement:

   1. Evidence for presence of malignant disease, inflammatory lesions, and/or vasculitis on cerebral magnetic resonance imaging (MRI)
   2. Infiltration of the cerebrospinal fluid by malignant B-cells, confirmed by lumbar puncture
7. History of or current relevant CNS pathology as epilepsy, seizure, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis
8. Cancer chemotherapy within 4 weeks prior to start of AFM11 treatment, or at least 4 times the respective half-lives, whichever is longer
9. Therapy with antibody, or antibody constructs within 4 weeks prior to the start of AFM11 treatment, or at least 4 half-lives, whichever is longer
10. Treatment with any investigational agent within 4 weeks prior to start of AFM11 treatment, or at least 4 times the respective half-life, whichever is longer
11. Contraindication for any of the concomitant medications
12. Abnormal renal or hepatic function as follows: aspartate aminotransferase (AST or SGOT) and/or alanine aminotransferase (ALT or SGPT) ≥ 2.5 × ULN; total bilirubin ≥ 1.5 × ULN; serum creatinine ≥ 2 × ULN; creatinine clearance < 50 mL/minute
13. History of malignancy other than B-cell lymphoma or B-precursor ALL within 5 years prior to study entry, with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix
14. Uncontrolled infections; known bacteremia
15. Any concurrent disease or medical condition that is deemed to interfere with the conduct of the study as judged by the Investigator
16. Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), high risk of or known uncontrolled arrhythmia
17. Regular dose of corticosteroids during the 4 weeks prior to start of AFM11 treatment of this study or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent, or any other immunosuppressive therapy within 4 weeks prior to study entry. Exception is the pre treatment of rapidly progressing disease
18. Known infection with human immunodeficiency virus or chronic or acute infection with hepatitis B or hepatitis C virus
19. Pregnant or nursing women or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 3 months thereafter. Male patients not willing to ensure that during the study and at least 3 months thereafter no fathering takes place. Effective methods of contraception include intrauterine device (IUD), combined (estrogen- and progesterone-containing) hormonal contraception (oral, vaginal ring or transdermal patch) with an ethinylestradiol dose of at least 30 µg, plus use of male condoms (preferably with spermicides), female condoms, a female diaphragm, or a cervical cap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious and non-serious adverse events as a measure of safety and tolerability of increasing doses and different infusion times of AFM11 | From first administration of continuous infusion over 2 weeks in step 1 (or 4 weeks in step 2) followed by 2 weeks of treatment break
  Measure of occurence of adverse events (AEs), laboratory testing (chemistry and hematology), physical examination, vital signs, cardiac monitoring, and neurological assessments

SECONDARY OUTCOMES:
Maximum Plasma Concentration of AFM11 (Cmax) | Multiple time points during the 2 weeks of treatment in step 1 and 4 weeks of treatment in step 2
  The maximum observed concentration of AFM11 in plasma will be determined.
Area Under the Curve (AUC) | Prior to initial dose on Day 1 and at multiple time points during the 2 weeks of treatment in step 1 and 4 weeks of treatment in step 2
  The area under the concentration versus time curve from time zero to the sampling time will be determined.
Clinical efficacy of AFM11 in ALL | Baseline and after treatment (week 3 in step 1 or week 4 in step 2)
  Measured by bone marrow assessment (complete response [CR], complete response with incomplete hematological recovery [CRh], and minimal residual disease [MRD])
Measurement of immunological markers | Prior to initial dose on Day 1 and at multiple time points during the 2 weeks of treatment in Step 1 and 4 weeks of treatment in Step 2
  Immunological markers like lymphocytes and cytokine levels in serum will be measured at different time points during the 4 weeks of treatment and 30 days thereafter to assess the level of activity resulting from administration of AFM11.

CONTACTS AND LOCATIONS:
Locations (12):
- Austria (3):
  - LKH-Universitätsklinikum Graz, Graz
  - Kepler Universitätsklinikum Linz, Linz
  - Uniklinikum Salzburg, Salzburg
- University Hospital, Brno, Czechia
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Poland (2):
  - Independent Public Healthcare Municipal Hospital, Chorzów
  - University Hospital, Krakow
- Russia (3):
  - Baranov Republican Hospital, Petrozavodsk
  - First Pavlov State Medical University, Saint Petersburg
  - Almazov NW Federal Medical Research Center, Saint Petersburg

REFERENCES:
- [Derived] Topp M, Dlugosz-Danecka M, Skotnicki AB, Salogub G, Viardot A, Klein AK, Hess G, Michel CS, Grosicki S, Gural A, Schwarz SE, Pietzko K, Gartner U, Strassz A, Alland L, Mayer J. Safety of AFM11 in the treatment of patients with B-cell malignancies: findings from two phase 1 studies. Trials. 2023 Jan 3;24(1):4. doi: 10.1186/s13063-022-06982-7. PMID 36597128